CLINICAL TRIAL: NCT02904434
Title: Gastrointestinal Implications of Voriconazole Exposure: Determining Age-dependent Differences in Intestinal Metabolism Affecting Oral Bioavailability of Voriconazole in Children
Brief Title: Gastrointestinal Implications of Voriconazole Exposure
Acronym: GIVE
Status: Withdrawn | Type: Observational
Why Stopped: IRB terminated the study
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 16-012970
Record Dates: First submitted 2016-09-07; First posted 2016-09-19 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Infection
Keywords: voriconazole; absorption; pharmacokinetic; grapefruit juice; bioavailability; intestinal first-pass metabolism; pharmacokinetics; intestinal
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be drawn during 12 hours following voriconazole administration. Samples will be analyzed for voriconazole concentrations.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Voriconazole: Children (2-17 years old) will receive oral voriconazole as prescribed by their physicians as standard of care for the duration of the study.
  Interventions: Other: Grapefruit Juice

INTERVENTIONS:
Other: Grapefruit Juice — On day 1 of the study, subjects will receive their standard voriconazole dose with no grapefruit juice. On day 2 of the study, subjects will receive approximately 240mL of reconstituted grapefruit juice by mouth or via nasogastric tube 30 minutes prior to receiving a scheduled dose of voriconazole. Blood samples will be collected during the 12 hours following voriconazole dosing on both days of the study.

SUMMARY:
Voriconazole has better response rates, improved survival and less adverse side effects compared to other drugs for the treatment of invasive fungal infections making it a desirable therapeutic option for children. However, dosing is unpredictable in children and this leads to therapeutic failure. This study aims to understand the physiological differences between children and adults that leads to therapeutic failure of voriconazole in children.

DETAILED DESCRIPTION:
Voriconazole clearance in children (2-12 years old) is 3-fold higher and bioavailability is one half of adult values. An important gap in knowledge exists that explain the mechanisms that result in higher clearance and lower bioavailability of voriconazole and places children at a substantial risk for sub-therapeutic concentrations and treatment failures. Preliminary data suggests that intestinal first-pass metabolism is responsible for the lower bioavailability in children, but not in adults. By inhibiting intestinal metabolism with grapefruit juice, the extent of the effect of intestinal first-pass metabolism on voriconazole pharmacokinetics can be determined. Inpatient children at the Children's Hospital of Philadelphia who are receiving oral voriconazole as standard of care will be enrolled in an open label, cross-over clinical trial to monitor plasma voriconazole levels after voriconazole administration with and without grapefruit juice to inhibit intestinal metabolism of voriconazole. The proposed research will elucidate the role of intestinal metabolism in the reduced oral bioavailability of voriconazole in children, which can be incorporated into a model simulation to guide accurate dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 2-17 years old
2. Receiving oral voriconazole as standard of care and at steady-state concentrations (defined as 72 hours from first-dose or 72 hours with no dose change)
3. Informed Consent/Assent when appropriate

Exclusion Criteria:

1. Allergy or inability to receive the slushy solution, which will be prepared using commercially available frozen grapefruit juice concentrate, cherry syrup, and Sprite.
2. Receiving tacrolimus and/or cyclosporine, which are affected by the furanocoumarins, during study period
3. Suspected or known hepatic dysfunction (defined as liver function tests measured at 3x upper limit of normal within the past 1 month, when measured as standard of care)
4. Receiving renal replacement therapy (example peritoneal dialysis, hemodialysis, continuous veno-venous hemofiltration, continuous veno-venous hemodialysis)
5. Receiving therapy with extracorporeal membrane oxygenation (ECMO)
6. Patients with documented pancytopenia, diarrhea, mucositis, or active infection

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children (2-17 years old) who are being treated at The Children's Hospital of Philadelphia and receiving oral voriconazole as standard of care will be eligible to enroll in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
VoriconazoleArea Under the Curve (AUC) | Two days
  Pharmacokinetic samples will be collected

SECONDARY OUTCOMES:
Voriconazole Apparent Bioavailability | Two days
  Pharmacokinetic samples will be collected
Voriconazole Apparent Clearance | Two days
  Pharmacokinetic samples will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Athena Zuppa, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No